CLINICAL TRIAL: NCT02331173
Title: Clinical Evaluation of Patients With X-linked Retinoschisis (XLRS)
Brief Title: Clinical Evaluation of Patients With X-linked Retinoschisis
Status: Completed | Type: Observational
Sponsor: Beacon Therapeutics (Industry)
Collaborators: Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Other Study IDs: XLRS-001
Record Dates: First submitted 2014-12-08; First posted 2015-01-06 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: X-linked Retinoschisis; XLRS
Keywords: XLRS; RS1; maculoschisis
MeSH Terms: conditions — Retinoschisis | interventions — dorzolamide; brinzolamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Main Study Group: All subjects enrolled in this study will be seen every 6 months following the screening visit. During the 3 main study visits, a series of tests will be performed to assess visual function. Some of these tests are part of routine care that patients would receive on an annual basis regardless of study participation. Other tests are being performed to determine if they are effective at monitoring disease progression in this population. For each of the 3 main study visits, testing may be spread over multiple days to ensure completion of all tests.
- Carbonic anhydrase inhibitor sub-study: Subjects with maculoschisis may be offered topical treatment with CAIs. These subjects will be asked to visit the study site at 1 month and 3 months after starting topical treatment. During these additional visits, subjects will undergo a dilated eye exam, BCVA, and SD-OCT imaging to assess efficacy of treatment (i.e. reduction of maculoschisis).
  Interventions: Drug: Dorzolamide 2% TID or brinzolamide 1% TID

INTERVENTIONS:
Drug: Dorzolamide 2% TID or brinzolamide 1% TID — Dosing of all medications will be based upon standard of care. Standard dosing for the treatment of pediatric and adult patients with XLRS is as follows:
  * Topical dorzolamide 2% three times per day
  * Topical brinzolamide 1% three times per day
  Groups: Carbonic anhydrase inhibitor sub-study

SUMMARY:
The purpose of this study is to evaluate subjects with X-linked retinoschisis in a clinical setting to collect data on disease progression.

DETAILED DESCRIPTION:
The objective of the study is to evaluate subjects with XLRS in a clinical setting and gather data on disease progression. The data from this study will enhance the understanding of the natural history of this rare disease and will facilitate appropriately powered safety studies in a future gene therapy trial in humans.

ELIGIBILITY:
Inclusion Criteria:

Main Study:

* Clinical diagnosis consistent with XLRS
* Documented disease causing RS1 mutation
* 7 years of age or older
* Able to provide informed consent/assent
* Male

CAI sub-study:

• Presence of maculoschisis

Exclusion Criteria:

Main Study:

• Other eye diseases that might affect the results (e.g. history of retinal detachment, glaucoma, cataracts that prohibit imaging, or any other eye pathology that in the opinion of the investigator would preclude enrollment)

CAI Sub-study:

Exclusion Criteria

* Already being treated with CAIs
* Previous documented failure to respond to CAI treatment

Any drug-specific contraindication/precaution listed below (from www.micromedex.com):

Topical Eye Drop Dorzolamide Hydrochloride

Contraindications:

• hypersensitivity to dorzolamide products, including sulfa allergies

Precautions:

* dorzolamide is a sulfonamide that is absorbed systemically, sulfonamide hypersensitivity reactions may occur
* angle-closure glaucoma
* concomitant use of oral carbonic-anhydrase inhibitors
* conjunctivitis and lid reactions reported with chronic administration
* moderate to severe renal (CrCl less than 30 mL/min) or hepatic insufficiency
* ocular infection or inflammation
* recent ocular surgery

Topical Eye Drop Brinzolamide

Contraindications:

• hypersensitivity to any component of the product, including sulfa allergies

Precautions:

* concomitant use of oral carbonic anhydrase inhibitors is not recommended
* contact lens use; remove contact lenses prior to administration, allow 15 minutes before reinsertion
* hypersensitivity to sulfonamides; severe reaction may occur; discontinue if signs or symptoms appear
* low corneal endothelial cell counts; increased risk of corneal edema
* renal impairment, severe (CrCl less than 30 mL/min); use not recommended

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential subjects will be identified from the Oregon Retinal Degeneration Center (ORDC) database and the Retina and Ophthalmic practices at Oregon Health and Science University Casey Eye Institute, Retina Foundation of the Southwest and Kellogg Eye Center.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Disease progression in subjects with XLRS | Every 6 months for 18 months

SECONDARY OUTCOMES:
Disease progression using microperimetry, a non-standard of care visual function test | Every 6 months for 18 months
Disease progression using electroretinograms (ERGs), a non-standard of care visual function test | Every 6 months for 18 months
Disease progression using the reading speed test, a non-standard of care visual function test | Every 6 months for 18 months
Disease progression using the contrast sensitivity test, a non-standard of care visual function test | Every 6 months for 18 months
Disease progression using a quality of life questionnaire | Every 6 months for 18 months
Change in maculoschisis while receiving carbonic anhydrase inhibitors | All study visits, Months 1, 3, 6, 12, and 18
Change in visual function while receiving carbonic anhydrase inhibitors | All study visits, Months 1, 3, 6, 12, and 18

CONTACTS AND LOCATIONS:
Overall Officials: Matt Feinsod, MD, Study Director — Applied Genetics Technologies Corporation
Locations (3):
- United States (3):
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Casey Eye Institute, Oregon Health and Sciences University, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas

REFERENCES:
- [Derived] Pennesi ME, Birch DG, Jayasundera KT, Parker M, Tan O, Gurses-Ozden R, Reichley C, Beasley KN, Yang P, Weleber RG, Bennett LD, Heckenlively JR, Kothapalli K, Chulay JD, For The Xlrs-Study Group. Prospective Evaluation of Patients With X-Linked Retinoschisis During 18 Months. Invest Ophthalmol Vis Sci. 2018 Dec 3;59(15):5941-5956. doi: 10.1167/iovs.18-24565. PMID 30551202